CLINICAL TRIAL: NCT04677062
Title: Safety, Galenic Acceptability and Efficacy of GV-328 Lozenges in Children With Oral Aphthosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Francisco Guinot-Jimeno, Jefe departamento de odontopedaitria, Universitat Internacional de Catalunya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UIC-ODP-VIÑAS
Record Dates: First submitted 2020-12-11; First posted 2020-12-21 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Aphthous Stomatitis
Keywords: aphthous lesion; hyaluronic acid
MeSH Terms: conditions — Stomatitis, Aphthous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GV-328 (Experimental): The treatment should be carried out for 4 days. Children between 3 and 6 years old had to consume 4 pills a day, children between 7 and 10 years old 5 pills, and children between 11 and 13 years old up to 6 pills. The patient had to slowly thin the tablet in the mouth, maintaining direct contact with the area to be treated.
  The study consisted of 2 visits, one initial and one final. In the initial visit , the documentation (informed consent) and the treatment were delivered. During this visit, baseline assessments of pain level, functional limitation, marginal mucosal edema, and lesion size were recorded. In addition, a photograph of the area to be treated was taken. Parents were also given a chart, in which they had to record the intensity of pain daily using the Wong-Baker face scale.
  Interventions: Drug: GV-328

INTERVENTIONS:
Drug: GV-328 — Patients with GV-328 treatment

SUMMARY:
The aim of the study was to assess the safety, acceptability, and efficacy of product GV-328 for the treatment of childhood oral aphthous lesion.

DETAILED DESCRIPTION:
Prospective study carried out in the Pediatric Dentistry Department of the International University of Catalonia. The sample was made up of children between 3 and 13 years old. Baseline pain status, functional limitation, edema and lesion diameter were evaluated. The treatment lasted 4 days. The parents recorded the intensity of the pain and the number of pills provided daily. Statistical significance was accepted with p≤0.05 and a 95% confidence interval.

A total sample of 33 patients, 11 boys (33 %) and 22 girls (67 %) was obtained. The average age of the children was 7.8 years (SD: 1.41). Numerical variables referring to pain, inflammation and edema presented statistically significant improvements (p-value <0.05). Healing efficacy was demonstrated in 13 cases (39 %) and only 3 cases (9 %) reported poor taste acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 3-13 years.
* Children who presented canker sores.

Exclusion Criteria:

* Patients who presented canker sores with 48 h of evolution.
* Patients with diabetic disorders.

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
The level of pain was measured on the Wong-Baker Faces Scale (WBFS) | 4 DAYS
  It consists of a 6-point scale that ranges from 0 (no pain) to 5 (excruciating pain).

SECONDARY OUTCOMES:
The degree of functional limitation and edema in the marginal mucosa were measured using a Likert scale. | 4 DAYS
  (0-absent, 1-mild, 2-moderate, 3-intense, 4-very intense).

OTHER OUTCOMES:
The baseline size of the main lesion was also classified according to its diameter | 4 DAYS
  <0.5 cm, 0.5-1.0cm or> 1.0 cm.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain